CLINICAL TRIAL: NCT01532154
Title: Fampridine Pregnancy Exposure Registry
Status: Terminated | Type: Observational
Why Stopped: Due to low enrollment, registration closed in agreement with the Regulatory Agency
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 218MS402
Record Dates: First submitted 2011-12-15; First posted 2012-02-14 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis; Pregnancy
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fampridine — As prescribed and taken after the last menstrual period prior to becoming pregnant or anytime during the pregnancy
  Other Names: dalfampridine; Ampyra; BIIB041; fampridine prolonged-release tablets; Fampyra

SUMMARY:
This is a global pregnancy registry to evaluate the outcomes of pregnancy in women with multiple sclerosis who have been exposed to prolonged-release fampridine since the first day of their last menstrual period prior to conception or at any time during pregnancy.

DETAILED DESCRIPTION:
There are no mandatory physician visits. The registry will collect pregnancy outcome data from the participants health care provider during the prenatal follow up (6-7 months gestation), pregnancy outcome (4 weeks after estimated delivery date) and finally the pediatric follow up (at 4 weeks and 12 weeks post birth).

ELIGIBILITY:
Key Inclusion Criteria:

* Documentation that the patient was exposed to prolonged-release fampridine since the first day of her last menstrual period (LMP) prior to conception or at any time during pregnancy. (If exposure dates are unknown, the reporter must be able to specify or estimate trimester of exposure.)
* The outcome of the pregnancy must not be known at the time of report.

Key Exclusion Criteria:

* None

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be pregnant female participants with multiple sclerosis who have been exposed to prolonged release fampridine since the first day of the last menstrual period or at any time during pregnancy. This information will be from ongoing fampridine clinical studies or the post-marketing setting. The outcome of the pregnancy must not be known at the time of report.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Spontaneous abortions | < 22 weeks of gestation
Elective or therapeutic terminations | Up to 9 months of pregnancy
Ectopic pregnancy | Up to 9 months of pregnancy
Fetal death including still births | >22 weeks of gestation or weighing 500 grams
Live born infants | During delivery time ( at expected average 9 months of pregnancy)
Premature births | Delivered before 37 Weeks of gestation
Maternal death | During pregnancy, labor or delivery
Neonatal death | Prior to 28 days of life
Birth Defects | Delivery time (expected 9 months of pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Hopital Pitie Salpetriere, Paris, France